CLINICAL TRIAL: NCT01368549
Title: Metanx® P.L.U.S. Program (Progress Through Learning, Understanding & Support)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pamlab, L.L.C. (Industry)
Collaborators: InfoMedics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Pamlab, Inc. (Industry)
Other Study IDs: M-005
Record Dates: First submitted 2011-05-17; First posted 2011-06-08 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Metanx; diabetes; neuropathy; folic acid; folate; L-methylfolate; vitamin B6; Pyridoxal 5'-phosphate; vitamin B12; methylcobalamin; DPN
MeSH Terms: conditions — Diabetes Mellitus | interventions — metanx

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Metanx®: Subjects with Diabetic Peripheral Neuropathy who have been prescribed Metanx® daily.
  Interventions: Other: Metanx® (a medical food)

INTERVENTIONS:
Other: Metanx® (a medical food) — Metanx® is an orally-administered medical food, and each tablet contains 3mg of L-methylfolate, 35mg of Pyridoxal-5'-phosphate, and 2 mg of Methylcobalamin- which are the biologically active and immediately bioavailable forms of folate, vitamin B6, and vitamin B12, respectively. Dosage will be 1 tablet BID.

SUMMARY:
This study will be an observational study in which patients who have been prescribed Metanx® are invited to participate in surveys regarding their experiences with Metanx®. The purpose of this study is to increase the understanding of the role of Metanx® in managing diabetic neuropathy, provide patients with personalized education and support, and contribute to the overall understanding of the needs and concerns of patients being treated for diabetic neuropathy.

DETAILED DESCRIPTION:
Surveys used to conduct this study will be administered via telephone or online by InfoMedics, Inc., a company with a system for developing such patient-physician feedback programs. Participating physicians will ask their patients to participate in the program after Metanx® has been prescribed and provide them with a brochure containing an introduction to the program and instructions on how to enroll. Patients self-enroll, take a brief survey before starting their Metanx® prescription, and then two brief follow-up surveys at 6 weeks and 12 weeks. As patients complete surveys within the study, their physician will receive individualized feedback reports outlining their patient's treatment experience and progress. Patients will also receive a copy of their own reports, to help encourage them to continue taking Metanx® as directed. Patients will also receive educational materials about managing their diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* New Metanx® Start
* Diagnosis of Diabetic Peripheral Neuropathy who have been prescribed Metanx® to help metabolic management of endothelial dysfunction.

Exclusion Criteria:

* Patients who do not meet ADA criteria for DPN diagnosis.
* If participant indicates that he or she did not get a prescription for Metanx®, he/she will not be able to complete the survey(s).
* For follow-up surveys, if the participant indicates that he/she has not been taking Metanx®, he/she will not be able to complete the survey(s).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Diabetic Peripheral Neuropathy Who Have Been Prescribed Metanx®
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
To determine if Metanx® improves neuropathic symptoms as evaluated by the Neuropathy Total Symptom Score-6 (NTSS-6) | Baseline, Week 6 and Week 12

SECONDARY OUTCOMES:
To determine if Metanx® affects a subject's pain level using a 10-point Visual Analog Scale (VAS) | Baseline, Week 6 and Week 12
To determine if Metanx® affects a subject's "quality of life" as determined by a symptom impact module. | Baseline, Week 6 and Week 12
To determine overall patient satisfaction with Metanx® using a 10-point satisfaction scale | Baseline, Week 6 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trippe, M.D., Principal Investigator — Endocrinology Associates
Locations (1):
- Endocrinology Associates, Montgomery, Alabama, United States